CLINICAL TRIAL: NCT05098483
Title: Clinical and Radiographic Evaluation of Regenerative Endodontics Using MTA and Biodentine for Non-vital Primary Molars Compared to Conventional Root Canal Treatment. (A Randomized Controlled Clinical Trial)
Brief Title: Regenerative Endodontics for Non-vital Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mai Hasaballah, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ain-Shams-University
Record Dates: First submitted 2021-09-17; First posted 2021-10-28 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2023-10

CONDITIONS: Pulp and Periapical Tissue Disease
Keywords: Regenerative endodontic treatment
MeSH Terms: interventions — Regeneration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional root canal treatment (Active Comparator): The caries will be removed. An excavator will be used to remove the coronal portion of the dental pulp while the radicular portion will be cleaned using k- files. 2.5% Sodium hypochlorite will be used as irrigant solution.The canals will be filled with ZOE cement and a stainless-steel crown will be inserted to restore the tooth.
  Interventions: Procedure: Conventional Root canal treatment in primary molars
- Regenerative endodontic treatment using MTA (Experimental): Access cavity will be prepared in each primary molar then each canal will be copiously irrigated by sodium hypochlorite. Triple antibiotic paste will be inserted in eash canal then sealed with temporary restoration till the second visit.
  In the second visit canals will be irrigated with EDTA, after that induction of bleeding will be created by overinstumentation inside each canal. Finally sealed with MTA under the GIC restoration and S.S.C
  Interventions: Procedure: Regeneration in primary molars by using MTA
- Regenerative endodontic treatment using Biodentine (Experimental): Access cavity will be prepared in each primary molar then canals will be copiously irrigated by sodium hypochlorite. Mixture of Triple antibiotic paste will be introduced in eash canal then cavity will be sealed with temporary restoration till the second visit.
  In the second visit canals will be irrigated with EDTA, after that bleeding will be created by overinstumentation inside each canal. Finally sealed with biodentine under the GIC restoration and S.S.C
  Interventions: Procedure: Regeneration in primary molars by using biodentine

INTERVENTIONS:
Procedure: Regeneration in primary molars by using MTA — Regenerative endodontic procedure in nonvital primary molars using MTA capping material
  Arms: Regenerative endodontic treatment using MTA
Procedure: Regeneration in primary molars by using biodentine — Regenerative endodontic treatment in primary molars with biodentine as capping material
  Arms: Regenerative endodontic treatment using Biodentine
Procedure: Conventional Root canal treatment in primary molars — Removal of pulp tissue from the canals of primary molars
  Arms: Conventional root canal treatment

SUMMARY:
Non-vital primary molars will be treated with regenerative endodontic idea using different capping materials aiming to replace the necrotic pulp tissue with biological one and to provide perfect seal over the scaffold

DETAILED DESCRIPTION:
Non-vital primary molars that fulfill the eligibility criteria will be randomly assigned into one of the 3 study groups:

Group 1: conventional root canal treatment Group 2: Regenerative endodontic treatment using MTA Group3: Regenerative endodontic treatment using Biodentine Each group will be followed up for 12 months

ELIGIBILITY:
Inclusion Criteria:

* Non-vital mandibular primary second molar.
* Restorable tooth

Exclusion Criteria:

* Patients allergic to medicaments or antibiotics necessary to complete the procedure.
* Special Health Care Needs
* Excessive mobility
* Presence of internal or external root resorption.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-10-26 (Actual); Study Completion 2024-10-26 (Actual)

PRIMARY OUTCOMES:
Clinical measures | 12 months
  39 children with no pain or swelling (i.e) successful outcomes
Radiographic measures | 12 months
  39 children with no furcal radiolucency or presence of internal resorption. (i.e) successful outcome

CONTACTS AND LOCATIONS:
Overall Officials: Mai Hasaballah, Principal Investigator — AinShams University
Locations (1):
- Mai Mahmoud Hasaballah, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No